CLINICAL TRIAL: NCT03253718
Title: Technical Development of Clinical Laboratory Studies
Status: Withdrawn | Type: Observational
Why Stopped: Study withdrawn due to limited personnel, time, resources.
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170150; 17-N-0150
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy Volunteers between 18 and 68 years of age

SUMMARY:
Background:

The Human Motor Control Section does tests for people with movement disorders. In order to be sure when a test is normal or abnormal, normal values must be determined in a large group of healthy volunteers (HVs). Therefore, the researchers want to study the techniques in HVs. They will use the results as the standard of comparison in future clinical studies.

Objective:

To get enough normal results in movement tests to use in clinical studies.

Eligibility:

Healthy adults ages 18-68

Design:

Participants will be screened with medical history and physical and neurological exams.

Participants will have 1 to 3 visits. They may have:

Small sticky electrodes attached to the skin on the hands/arms and neck. These will measure muscle activity.

Tiny shocks given to a finger. Participants will be asked if they felt 1 or 2 shocks. This will be done to each hand over about 30 minutes total.

A questionnaire about anxiety.

Acoustic startle reflex test. Small electrodes will be stuck to the eye, hand, and leg. Sensors will be stuck to the palms. Small metal electrodes on the chest and inner arm will measure heart rate. Participants will wear headphones. Once everything is in place, participants will hear a low sound for about 10 minutes. They will hear a short louder sound every 45 60 seconds.

DETAILED DESCRIPTION:
Objective

The purpose of this protocol is to get adequate normal values to compare in clinical patient studies.

Study population

There will be two techniques developed in this study: Somatosensory Temporal Discrimination Threshold (STDT) and Acoustic Startle Reflex (ASR). For both studies we will collect data systematically in an adequate sample of normal subjects.

We plan to recruit the following number of healthy volunteers (HV s) for each study.

STDT: 50 HV

ASR: 50 HV

Design

Subjects will come for up to 3 outpatient visits, during which they will participate in at least the STDT or the ASR. Before participation in any study, all participants will undergo screening for medical history and physical examination.

For the STDT, the index finger in both hands will be stimulated.

For the ASR, auditory stimulation will be administered at varying intervals. Subjects will also be asked to complete State Trait Anxiety Inventory (STAI) before participation in the study.

Outcome measures

STDT: discrimination threshold value

ASR: EMG response from seven muscles, heart rate, and galvanic skin response

ELIGIBILITY:
* INCLUSION CRITERIA:
* Between 18 and 68 years of age
* Ability to give informed consent
* Able to understand the procedures and requirements of the study

EXCLUSION CRITERIA:

* Diagnosis of a neurological disorder
* Illegal drug use within the past six months. The intent is to exclude those with drug use that may affect study results
* Self-reported consumption of >7 alcoholic drinks a week for women and >14 alcoholic drinks a week for men
* Unwillingness to abstain from caffeine or alcohol on the day of the study
* Abnormal findings on neurological exam of clinical significance
* History of or current brain tumor, stroke, head trauma with loss of consciousness > few seconds, epilepsy or seizures
* Open scalp wounds or scalp infections
* For ASR, unwillingness to abstain from the use of cigarettes on the day of the study

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HV s will be recruited through NIH Patient Recruitment and Public Liaison Office and from our database of individuals who have participated in prior studies and are interested in being contacted for additional studies.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
STDT values in both hands | throughout protocol
  Sub-study 1: Somatosensory Temporary Discrimination Threshold (STDT): STDT values in both hands.
The amount, latency and duration of muscle activity, heart rate, and skin conductance. | throughout protocol
  Sub-study 2: Acoustic Startle Reflex (ASR): The amount, latency and duration of muscle activity, heart rate, and skin conductance.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-N-0150.html